CLINICAL TRIAL: NCT01525602
Title: A Phase 1b Study to Assess the Safety of PLX3397 and Paclitaxel in Patients With Advanced Solid Tumors
Brief Title: Safety Study of PLX3397 and Paclitaxel in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Plexxikon (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLX108-07
Record Dates: First submitted 2012-01-31; First posted 2012-02-03 (Estimated); Results first posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Solid Tumors
Keywords: advanced, incurable solid tumors
MeSH Terms: interventions — pexidartinib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 (Experimental): Open-label, sequential PLX3397 single-agent dose escalation in combination with paclitaxel in approximately 30 patients with advanced solid tumors. Enrollment completed.
  (Closed to recruitment)
  Interventions: Drug: PLX3397; Drug: Paclitaxel
- Part 2 (Experimental): Extension cohort at the RP2D of single-agent PLX3397 in combination with paclitaxel in approximately 30 patients in advanced solid tumors. Enrollment completed.
  (Closed to recruitment)
  Interventions: Drug: PLX3397; Drug: Paclitaxel
- Part 3 (Experimental): Extension cohort at the RP2D of single-agent PLX3397 in combination with paclitaxel in approximately 30 patients with advanced, metastatic, or non-resectable, platinum-resistant or -refractory epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer.
  (Closed to recruitment)
  Interventions: Drug: PLX3397; Drug: Paclitaxel

INTERVENTIONS:
Drug: PLX3397 — PLX3397 tablets, 200mg
  Other Names: Pexidartinib
Drug: Paclitaxel — Paclitaxel IV
  Other Names: Onxol

SUMMARY:
This was a 3-part study designed to explore the safety and tolerability of escalating doses of PLX3397 with weekly paclitaxel to establish a recommended Phase 2 dose (RP2D), to confirm RP2D in participants with advanced non-resectable solid tumors, and to determine the efficacy of PLX3397 600 mg twice daily (BID) administered in combination with weekly paclitaxel in participants with advanced, metastatic or non-resectable, platinum-resistant or -refractory epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with:

  * Part 1 (enrollment closed): an advanced, incurable solid tumor
  * Part 2 (enrollment closed): an advanced, incurable solid tumor for whom a taxane would be considered a reasonable chemotherapy option
  * Part 3 (enrollment closed): advanced, metastatic or non-resectable epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer with

    * platinum-resistant cancer, defined as disease that responded to a platinum-containing chemotherapy regimen, but demonstrated recurrence within six months following the completion of that platinum-containing regimen, OR
    * platinum-refractory cancer, defined as disease failed to achieve at least a partial response to a platinum-containing regimen (i.e., stable disease or actual disease progression), AND
    * have not been treated with a taxane within six months of Cycle 1 Day 1 (C1D1), AND
    * have not been treated with weekly paclitaxel after first-line treatment in which weekly paclitaxel plus a platinum is permitted
* Part 3: Patients must have target (≥2 cm diameter) or non-target lesion cancer that is accessible for core biopsies before starting on study and after one cycle of treatment.
* Patients with stable brain metastases are eligible for this trial. However, patients must not have required steroid treatment for their brain metastases within 30 days of Screening.
* Bone-directed therapy (e.g., bisphosphonates or denosumab) is permitted.
* Washout from any prior investigational therapy of at least five times the T1/2 prior to C1D1
* Washout from any prior biologic or targeted therapy at least 4 weeks or five times the plasma half-life (T1/2) (whichever is shorter) prior to C1D1
* Washout from prior chemotherapy of at least 2 weeks or 1 elimination half-life, whichever is longer, prior to C1D1
* Washout from prior hormonal therapy of at least 2 weeks prior to C1D1
* Washout of at least 2 weeks from the most recent radiation treatment prior to C1D1
* Resolution of all prior treatment-related toxicities to Grade 1 or less, except for Grade 2 fatigue or alopecia prior to C1D1
* Age eighteen years or older
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2, inclusive
* Anticipated life expectancy of at least 12 weeks
* Adequate bone marrow reserve: absolute neutrophil count (ANC) ≥1500/mm3, platelets ≥100,000/mm3
* Adequate renal function: serum creatinine <1.5 x ULN or calculated creatinine clearance (CrCl) >60 mL/min using Cockcroft-Gault formula
* Adequate hepatic function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2.5 x upper limit of normal (ULN), Total and Direct Bilirubin <1.5 x ULN. However, in the presence of liver metastases, AST and ALT must be <5 x ULN
* Cardiac ejection fraction ≥50%, and QT interval corrected by Fridericia's formula (QTcF) <450 ms (males) or <470 ms (females) on electrocardiogram (ECG) at Baseline.
* Able to swallow capsules and maintain adequate hydration
* Ability to give written informed consent and willing to comply with the requirements of the protocol; and for Part 3, to give written informed consent for 2 cancer biopsy procedures
* Women of child-bearing potential must agree to use an effective method of birth control during treatment and for three months after receiving their last dose of study drug. Fertile men must also agree to use an acceptable method of birth control while on study drug and for at least 3 months after last dose.

Exclusion Criteria:

* Presence of an active secondary malignancy.

  * Patients with a non-melanomatous, in situ malignancy or disease that is completely resectable with surgery may be considered after discussion with the Medical Monitor
  * Patients with a completely treated prior malignancy with no evidence of disease for ≥3 years are eligible
* Refractory nausea and vomiting, malabsorption, external biliary shunt or significant small bowel resection that would preclude adequate absorption of PLX3397
* Ongoing treatment with any other investigational therapy
* Prior anaphylactic or severe hypersensitivity reaction to paclitaxel or Cremophor-containing agent.
* Persistent grade 2 fatigue at Baseline.
* Severe, concurrent illness including congestive heart failure, significant cardiac disease and uncontrolled hypertension, that would likely prevent the patient from being able to comply with the study protocol
* Active untreated infection
* Known chronic active Hepatitis B or C, or HIV infection
* The presence of a medical or psychiatric condition that, in the opinion of the Principal Investigator, makes the patient inappropriate for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-05; Primary Completion 2017-12 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Univeristy of California, San Francisco, San Francisco, California
  - University of Colorado, Anschutz Cancer Pavilion, Aurora, Colorado
  - Sylvester Comprehensive Cancer Center/UMHC, Miami, Florida
  - Mayo Clinic, Rochester, Minnesota
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 74 participants (54 in Parts 1 and 2; 20 in Part 3) who met all inclusion and none of the exclusion criteria were enrolled in this study.
Pre-assignment Details: An open-label study. In Part 1 (dose escalation), participants were sequentially enrolled and received doses of PLX3397 600 to 1600 mg/day. In Part 2 (dose expansion), PLX3397 was administered at the recommended phase 2 dose with paclitaxel. In Part 3, PLX3397 was administered at 600 mg twice daily with paclitaxel; 2 participants were not dosed.
Groups:
- Part 1: Cohort 1; 600 mg/Day: Participants with advanced solid tumors who received PLX3397 600 mg/day.
- Part 1: Cohort 2; 800 mg/Day: Participants with advanced solid tumors who received PLX3397 800 mg/day.
- Part 1: Cohort 3; 1000 mg/Day: Participants with advanced solid tumors who received PLX3397 1000 mg/day.
- Part 1: Cohort 4; 1200 mg/Day: Participants with advanced solid tumors who received PLX3397 1200 mg/day.
- Part 1 and 2: Cohort 5; 1600 mg/Day: Participants with advanced solid tumors who received PLX3397 1600 mg/day.
- Part 3: PLX3397 600 mg BID: All participants with advanced solid tumors who received PLX3397 600 mg twice daily (BID) as Cycle 1 lead-in treatment. After Cycle 1, participants were treated with PLX3397 600 mg BID and paclitaxel 80 mg/m^2 IV weekly.
- Part 3: Paclitaxel 80 mg/m^2: All participants with advanced solid tumors who received paclitaxel 80 mg/m^2 intravenous weekly as Cycle 1 lead-in treatment. After Cycle 1, participants were treated with PLX3397 600 mg twice daily (BID) and paclitaxel 80 mg/m^2 IV weekly.
- Part 3: PLX3397 600 mg + Paclitaxel 80 mg/m^2: All participants who received PLX3397 600 mg twice daily (BID) + paclitaxel 80 mg/m^2 intravenous weekly as Cycle 1 lead-in treatment.
Period: Overall Study
Arm/Group | Part 1: Cohort 1; 600 mg/Day | Part 1: Cohort 2; 800 mg/Day | Part 1: Cohort 3; 1000 mg/Day | Part 1: Cohort 4; 1200 mg/Day | Part 1 and 2: Cohort 5; 1600 mg/Day | Part 3: PLX3397 600 mg BID | Part 3: Paclitaxel 80 mg/m^2 | Part 3: PLX3397 600 mg + Paclitaxel 80 mg/m^2
Started | 9 | 3 | 3 | 6 | 33 | 7 | 6 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 9 | 3 | 3 | 6 | 33 | 7 | 6 | 7
Not completed — Adverse Event | 1 | 0 | 1 | 1 | 3 | 3 | 0 | 1
Not completed — Disease progression | 6 | 3 | 2 | 5 | 22 | 2 | 3 | 3
Not completed — Clinical progression | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Non-compliance | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Unqualified based on biopsy; not dosed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants who were treated and included in the Safety Population (n=72).
Groups:
- Part 3: PLX3397 600 mg BID: All participants with advanced solid tumors who received PLX3397 600 mg BID as Cycle 1 lead-in treatment. After Cycle 1, participants were treated with PLX3397 600 mg BID and paclitaxel 80 mg/m^2 IV weekly.
- Part 3: Paclitaxel 80 mg/m^2: All participants with advanced solid tumors who received paclitaxel 80 mg/m^2 intravenous weekly as Cycle 1 lead-in treatment. After Cycle 1, participants were treated with PLX3397 600 mg BID and paclitaxel 80 mg/m^2 IV weekly.
- Part 3: PLX3397 600 mg + Paclitaxel 80 mg/m^2: All participants who received PLX3397 600 mg BID + paclitaxel 80 mg/m^2 intravenous weekly as Cycle 1 lead-in treatment.
- Total: Total of all reporting groups
Arm/Group | Part 1: Cohort 1; 600 mg/Day | Part 1: Cohort 2; 800 mg/Day | Part 1: Cohort 3; 1000 mg/Day | Part 1: Cohort 4; 1200 mg/Day | Part 1 and 2: Cohort 5; 1600 mg/Day | Part 3: PLX3397 600 mg BID | Part 3: Paclitaxel 80 mg/m^2 | Part 3: PLX3397 600 mg + Paclitaxel 80 mg/m^2 | Total
Number analyzed (Participants) | 9 | 3 | 3 | 6 | 33 | 7 | 5 | 6 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (14.2) | 55.0 (5.3) | 60.3 (11.1) | 58.7 (16.4) | 58.9 (10.7) | 64.0 (10.4) | 64.8 (4.9) | 59.7 (8.8) | 59.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 1 | 3 | 20 | 7 | 5 | 6 | 51
  Male | 3 | 0 | 2 | 3 | 13 | 0 | 0 | 0 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 4
  White | 9 | 2 | 3 | 5 | 29 | 7 | 5 | 5 | 65
  More than one race | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 3 | 3 | 6 | 33 | 7 | 5 | 6 | 72

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (>10%) Classified by Preferred Term Following PLX3397 Administered in Combination With Paclitaxel (Parts 1 and 2) (Safety Population)
Description: Treatment-emergent adverse events (TEAEs) reported by >10% of all participants in Parts 1 and 2 are reported.
Time Frame: From post first dose up to 28 days after the last dose, up to 5 years 9 months
Population: Safety events were assessed in the Safety Population.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Cohort 1; 600 mg/Day | Part 1: Cohort 2; 800 mg/Day | Part 1: Cohort 3; 1000 mg/Day | Part 1: Cohort 4; 1200 mg/Day | Part 1 and 2: Cohort 5; 1600 mg/Day
Number analyzed (Participants) | 9 | 3 | 3 | 6 | 33
percentage of participants
  Any TEAE | 100 | 100 | 100 | 100 | 100
  Gastrointestinal disorders | 89 | 67 | 100 | 83 | 91
  Nausea | 44 | 33 | 67 | 67 | 42
  Diarrhea | 33 | 33 | 67 | 50 | 39
  Vomiting | 33 | 0 | 33 | 33 | 36
  Constipation | 33 | 0 | 33 | 0 | 21
  General disorders/administrative site conditions | 89 | 100 | 67 | 100 | 79
  Fatigue | 78 | 100 | 33 | 83 | 70
  Edema peripheral | 11 | 33 | 0 | 33 | 27
  Pyrexia | 22 | 0 | 33 | 17 | 18
  Blood and lymphatic disorders | 89 | 100 | 67 | 50 | 73
  Anemia | 78 | 67 | 33 | 33 | 67
  Neutropenia | 22 | 33 | 33 | 33 | 12
  Metabolism and nutrition disorders | 78 | 67 | 33 | 83 | 67
  Decreased appetite | 78 | 33 | 0 | 67 | 36
  Hypokalemia | 22 | 33 | 0 | 33 | 27
  Hypophosphatemia | 11 | 33 | 0 | 17 | 24
  Skin and subcutaneous disorders | 56 | 100 | 100 | 100 | 55
  Alopecia | 11 | 33 | 33 | 67 | 24
  Rash | 11 | 33 | 33 | 0 | 27
  Pruritus | 0 | 33 | 0 | 17 | 15
  Respiratory, thoracic, and mediastinal disorders | 33 | 67 | 100 | 50 | 61
  Dyspnea | 22 | 33 | 0 | 50 | 33
  Cough | 11 | 0 | 0 | 33 | 18
  Investigations | 11 | 67 | 100 | 67 | 61
  Aspartate aminotransferase increased | 0 | 67 | 33 | 33 | 42
  Lymphocyte count decreased | 11 | 67 | 33 | 33 | 36
  White blood cell count decreased | 0 | 67 | 33 | 50 | 36
  Blood creatinine phosphokinase increased | 0 | 33 | 67 | 17 | 39
  Neutrohil count decreased | 0 | 33 | 0 | 17 | 36
  Alanine aminotransferase increased | 0 | 33 | 33 | 17 | 21
  Blood alkaline phosphatase increased | 0 | 33 | 33 | 17 | 21
  Respiratory rate increased | 0 | 0 | 33 | 17 | 12
  Weight decreased | 11 | 33 | 33 | 17 | 6
  Nervous system disorders | 44 | 67 | 67 | 67 | 55
  Dysgeusia | 11 | 0 | 33 | 50 | 36
  Dizziness | 33 | 0 | 0 | 17 | 12
  Neuropathy peripheral | 22 | 0 | 33 | 17 | 12
  Headache | 0 | 33 | 0 | 17 | 12
  Vascular disorders | 11 | 67 | 0 | 50 | 39
  Hypertension | 11 | 67 | 0 | 50 | 30
  Eye disorders | 11 | 67 | 33 | 33 | 30
  Periorbital edema | 0 | 33 | 33 | 0 | 15
  Vision blurred | 0 | 0 | 0 | 17 | 15
  Psychiatric disorders | 11 | 0 | 0 | 17 | 21
  Insomnia | 11 | 0 | 0 | 0 | 15

2. Primary Outcome: Percentage of Participants With TEAEs (>10%) Classified by Preferred Term Following PLX3397 Administered in Combination With Paclitaxel (Part 3) (Safety Population)
Description: Treatment-emergent adverse events (TEAEs) reported by >10% of all participants in Part 3 are reported.
Time Frame: From post first dose up to 28 days after the last dose, up to 5 years 9 months
Population: Safety events were assessed in the Safety Population.
Measure: Number; unit: percentage of participants
Arm/Group | Part 3: PLX3397 600 mg BID | Part 3: Paclitaxel 80 mg/m^2 | Part 3: PLX3397 600 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 7 | 5 | 6
percentage of participants
  Any TEAE | 100 | 100 | 100
  Gastrointestinal disorders | 100 | 100 | 83.3
  Nausea | 71.4 | 60 | 66.7
  Diarrhea | 57.1 | 40 | 50
  Constipation | 28.6 | 60 | 16.7
  Vomiting | 14.3 | 40 | 50
  Abdominal distension | 14.3 | 40 | 16.7
  Abdominal pain | 28.6 | 20 | 16.7
  Stomatitis | 0 | 40 | 16.7
  Colitis | 14.3 | 0 | 16.7
  Toothache | 14.3 | 20 | 0
  General disorders/administrative site conditions | 42.9 | 100 | 100
  Fatigue | 42.9 | 80 | 100
  Chills | 0 | 0 | 66.7
  Edema peripheral | 14.3 | 40 | 0
  Pyrexia | 0 | 0 | 50
  Chest pain | 14.3 | 20 | 0
  Face edema | 0 | 20 | 16.7
  Nervous system disorders | 57.1 | 100 | 66.7
  Dysgeusia | 42.9 | 40 | 33.3
  Neuropathy peripheral | 28.6 | 60 | 16.7
  Dizziness | 28.6 | 20 | 33.3
  Headache | 14.3 | 20 | 16.7
  Skin and subcutaneous tissue disorders | 57.1 | 80 | 50
  Alopecia | 42.9 | 80 | 16.7
  Pruritus | 14.3 | 20 | 16.7
  Rash | 0 | 40 | 0
  Respiratory, thoracic, and mediastinal disorders | 28.6 | 80 | 66.7
  Dyspnea | 28.6 | 40 | 33.3
  Epistaxis | 14.3 | 40 | 16.7
  Cough | 14.3 | 40 | 0
  Oropharyngeal pain | 14.3 | 20 | 0
  Musculoskeletal and connective tissue disorders | 28.6 | 60 | 66.7
  Pain in extremity | 14.3 | 20 | 33.3
  Myalgia | 0 | 0 | 33.3
  Investigations | 42.9 | 20 | 66.7
  Alanine aminotransferase increased | 14.3 | 20 | 16.7
  Aspartate aminotransferase increased | 14.3 | 20 | 16.7
  Blood bilirubin increased | 14.3 | 0 | 16.7
  Lymphocyte count decreased | 14.3 | 0 | 16.7
  Neutrophil count decreased | 0 | 0 | 33.3
  Metabolism and nutrition disorders | 42.9 | 60 | 33.3
  Decreased appetite | 42.9 | 60 | 16.7
  Blood and lymphatic system disorders | 28.6 | 40 | 50
  Anemia | 28.6 | 20 | 33.3
  Neutropenia | 0 | 20 | 16.7
  Infections and infestations | 28.6 | 20 | 50
  Pneumonia | 28.6 | 20 | 0
  Renal and urinary disorders | 28.6 | 0 | 50
  Dysuria | 14.3 | 0 | 16.7
  Urinary incontinence | 14.3 | 0 | 16.7
  Vascular disorders | 0 | 20 | 50
  Hypertension | 0 | 0 | 50
  Injury, poisoning, and procedural complications | 14.3 | 0 | 33.3
  Contusion | 14.3 | 0 | 16.7
  Reproductive system and breast disorders | 28.6 | 20 | 0
  Vaginal hemorrhage | 14.3 | 20 | 0

3. Primary Outcome: Best Overall Tumor Response Based on RECIST V1.1 Following PLX3397 Administered in Combination With Paclitaxel (Parts 1 and 2) (Efficacy Evaluable Population)
Description: Best overall tumor response (complete response [CR], partial response [PR], stable disease [SD], progressive disease [PD]) is reported, including participants who were not evaluable (NE). RECIST v1.1 for target lesions are assessed by magnetic resonance imaging, computed tomography, or positron emission tomography-computed tomography and are summarized as: CR, Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm; PR, At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; PD, at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (includes the baseline sum). In addition, the sum must also demonstrate an absolute increase of at least 5 mm; SD, Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: From post first dose up to 5 years 9 months post dose
Population: Best overall tumor response was assessed in the Efficacy Evaluable Population.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Cohort 1; 600 mg/Day | Part 1: Cohort 2; 800 mg/Day | Part 1: Cohort 3; 1000 mg/Day | Part 1: Cohort 4; 1200 mg/Day | Part 1 and 2: Cohort 5; 1600 mg/Day
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 20
percentage of participants
  Complete response (CR) | 0 | 0 | 0 | 0 | 5
  Partial response (PR) | 17 | 0 | 33 | 17 | 10
  Stable disease | 33 | 33 | 33 | 50 | 30
  Progressive disease | 50 | 67 | 33 | 33 | 45
  Unable to assess | 0 | 0 | 0 | 0 | 10
  Best overall response rate (CR or PR) | 17 | 0 | 33 | 17 | 15
  Clinical benefit rate (CR, PR, or stable disease) | 50 | 33 | 67 | 67 | 45

4. Primary Outcome: Best Overall Tumor Response Based on RECIST V1.1 Following PLX3397 Administered in Combination With Paclitaxel (Part 3) (Efficacy Evaluable Population)
Description: as for outcome 3
Time Frame: From 26 days (CR and PR) and 54 days (SD) up to 5 years 9 months post dose
Population: Best overall tumor response was assessed in the Efficacy Evaluable Population.
Measure: Number; unit: percentage of participants
Groups:
- Part 3: PLX3397 600 mg BID + Paclitaxel 80 mg/m^2: All participants who received PLX3397 600 mg BID + paclitaxel 80 mg/m^2 intravenous weekly as Cycle 1 lead-in treatment.
Arm/Group | Part 3: PLX3397 600 mg BID | Part 3: Paclitaxel 80 mg/m^2 | Part 3: PLX3397 600 mg BID + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 4 | 5 | 5
percentage of participants
  Complete response (CR) | 0 | 0 | 0
  Partial response (PR) | 0 | 40 | 20
  Stable disease (SD) | 50 | 0 | 20
  Progressive disease (PD) | 50 | 60 | 60
  Best overall response rate (CR or PR) | 0 | 40 | 20
  Clinical benefit rate (CR, PR, or stable disease) | 50 | 40 | 40

5. Secondary Outcome: Duration of Response Following PLX3397 Administered in Combination With Paclitaxel (Parts 1 and 2) (Efficacy Evaluable Population)
Time Frame: From the date of initial response until disease progression or death, whichever occurs first, up to 5 years 9 months post dose
Population: Duration of response was assessed in the Efficacy Evaluable Population.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Part 1: Cohort 1; 600 mg/Day | Part 1: Cohort 2; 800 mg/Day | Part 1: Cohort 3; 1000 mg/Day | Part 1: Cohort 4; 1200 mg/Day | Part 1 and 2: Cohort 5; 1600 mg/Day
Number analyzed (Participants) | 1 | 0 | 1 | 1 | 3
days | 171 (0) |  | 9 (0) | 66 (0) | 113.3 (68.8)

6. Secondary Outcome: Duration of Response Following PLX3397 Administered in Combination With Paclitaxel (Part 3) (Efficacy Evaluable Population)
Time Frame: as for outcome 5
Population: Duration of response based on patients with CR or PR was assessed in the Efficacy Evaluable Population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 3: PLX3397 600 mg BID | Part 3: Paclitaxel 80 mg/m^2 | Part 3: PLX3397 600 mg BID + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 0 | 2 | 1
days |  | 119 [NA to NA] — There were not enough events to estimate confidence intervals for the median duration of response. | 114 [NA to NA] — There were not enough events to estimate confidence intervals for the median duration of response.

7. Secondary Outcome: Progression-free Survival Following PLX3397 Administered in Combination With Paclitaxel (Part 3) (Efficacy Evaluable Population)
Description: Progression-free survival (PFS) is defined as the number of days from the start of therapy (i.e. Cycle 1 Day 1) to the date of first documented disease progression/relapse or death, whichever occurs first. If the disease progression/relapse does not occur, PFS will be censored as of the date of their last evaluable tumor assessments.
Time Frame: From the first day of treatment to the first documented disease progression or date of death, whichever occurred first, up to 5 years 9 months post dose
Population: Progression-free survival was assessed in the Efficacy Evaluable Population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 3: PLX3397 600 mg BID | Part 3: Paclitaxel 80 mg/m^2 | Part 3: PLX3397 600 mg BID + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 4 | 5 | 5
days | 117 [22 to 176] | 59 [44 to 175] | 56 [8 to 220]

8. Secondary Outcome: A Summary of Pharmacokinetic Parameter (Tmax) Following Exposure to PLX3397 (Parts 1 and 3)
Time Frame: Cycle 1, Day 15
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Groups:
- Part 1: 600 mg BID: Participants with advanced solid tumors who received PLX3397 600 mg BID administered as three 100-mg capsules in the morning and evening, or two 200-mg capsules in the morning and one 200-mg capsule in the evening.
- Part 1: 800 mg (400 mg BID): Participants with advanced solid tumors who received PLX3397 800 mg administered 400 mg BID.
- Part 1: 1000 mg (BID): Participants with advanced solid tumors who received PLX3397 1000 mg BID administered as five 100-mg capsules in the morning and evening, or three 200-mg capsules in the morning and two 200-mg capsules in the evening.
- Part 1: 1200 mg (600 mg BID); Part 3: 1200 mg (600 mg BID): Participants with advanced solid tumors who received PLX3397 1200 mg administered 600 mg BID.
- Part 1 and 2: 1600 mg (800 mg BID): Participants with advanced solid tumors who received PLX3397 1600 mg administered 800 mg BID.
Arm/Group | Part 1: 600 mg BID | Part 1: 800 mg (400 mg BID) | Part 1: 1000 mg (BID) | Part 1: 1200 mg (600 mg BID) | Part 1 and 2: 1600 mg (800 mg BID) | Part 3: 1200 mg (600 mg BID)
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 6 | 6
hours | 0 [0 to 4] | 2 [0 to 4] | 0 [0 to 4] | 2 [2 to 4] | 2 [2 to 4] | 2 [2 to 4]

9. Secondary Outcome: A Summary of Pharmacokinetic Parameter (Cmax) Following Exposure to PLX3397 (Parts 1 and 3)
Time Frame: Cycle 1, Day 15
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: 600 mg BID | Part 1: 800 mg (400 mg BID) | Part 1: 1000 mg (BID) | Part 1: 1200 mg (600 mg BID) | Part 1 and 2: 1600 mg (800 mg BID) | Part 3: 1200 mg (600 mg BID)
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 6 | 6
ng/mL | 3420 (41.4) | 6640 (26.5) | 4340 (27.6) | 8190 (39.6) | 8000 (50.5) | 8540 (17.8)

10. Secondary Outcome: A Summary of Pharmacokinetic Parameters (AUC[0-4h], AUC[0-6h], and AUC[0-12h]) Following Exposure to PLX3397 (Parts 1 and 3)
Time Frame: Cycle 1, Day 15
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set, except for AUC(0-6) which was not performed for Part 1 and 2 participants, only participants in Part 3.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1: 600 mg BID | Part 1: 800 mg (400 mg BID) | Part 1: 1000 mg (BID) | Part 1: 1200 mg (600 mg BID) | Part 1 and 2: 1600 mg (800 mg BID) | Part 3: 1200 mg (600 mg BID)
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 6 | 6
h*ng/mL
  AUC (0-4) | 12400 (41.0) | 21700 (25.7) | 13100 (38.6) | 28000 (34.5) | 26500 (46.5) | 27800 (17.5)
  AUC (0-6): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6
  AUC (0-6) |  |  |  |  |  | 40100 (19.4)
  AUC (0-12) | 36900 (37.1) | 59300 (16.0) | 44400 (30.7) | 75600 (34.2) | 70500 (36.7) | 71700 (21.2)

11. Secondary Outcome: Percentage of Participants With PLX3397-Related Treatment-emergent Adverse Events (>10%) by Preferred Term (Parts 1 and 2) (Safety Analysis Set)
Time Frame: From post first dose up to 28 days after the last dose, up to 5 years 9 months
Population: Safety events were assessed in the Safety Analysis Set.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Cohort 1; 600 mg/Day | Part 1: Cohort 2; 800 mg/Day | Part 1: Cohort 3; 1000 mg/Day | Part 1: Cohort 4; 1200 mg/Day | Part 1 and 2: Cohort 5; 1600 mg/Day
Number analyzed (Participants) | 9 | 3 | 3 | 6 | 33
percentage of participants
  Any Paclitaxel-related TEAE | 89 | 100 | 100 | 100 | 94
  Nausea | 22 | 33 | 33 | 50 | 36
  Diarrhea | 22 | 33 | 67 | 50 | 24
  Vomiting | 22 | 0 | 33 | 33 | 27
  Fatigue | 33 | 100 | 33 | 83 | 64
  Pyrexia | 11 | 0 | 33 | 0 | 12
  Anemia | 33 | 67 | 0 | 17 | 36
  Decreased appetite | 33 | 33 | 0 | 66 | 24
  Hypophosphatemia | 11 | 33 | 0 | 17 | 15
  Rash | 11 | 0 | 33 | 0 | 27
  Pruritus | 0 | 33 | 0 | 17 | 15
  Aspartate aminotransferase increased | 0 | 67 | 33 | 33 | 42
  White blood cell count decreased | 0 | 33 | 33 | 50 | 33
  Blood creatinine phosphokinase increased | 0 | 33 | 67 | 17 | 39
  Neutrophil count decreased | 0 | 33 | 0 | 17 | 21
  Alanine aminotransferase increased | 0 | 33 | 33 | 17 | 21
  Blood alkaline phosphatase increased | 0 | 33 | 33 | 17 | 18
  Dysgeusia | 0 | 0 | 33 | 67 | 30
  Hypertension | 11 | 67 | 0 | 50 | 21
  Periorbital edema | 0 | 33 | 33 | 0 | 15

12. Secondary Outcome: Percentage of Participants With Paclitaxel-Related Treatment-emergent Adverse Events (>10%) by Preferred Term (Parts 1 and 2) (Safety Analysis Set)
Time Frame: From post first dose up to 28 days after the last dose, up to 5 years 9 months
Population: Safety events were assessed in the Safety Analysis Set.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Cohort 1; 600 mg/Day | Part 1: Cohort 2; 800 mg/Day | Part 1: Cohort 3; 1000 mg/Day | Part 1: Cohort 4; 1200 mg/Day | Part 1 and 2: Cohort 5; 1600 mg/Day
Number analyzed (Participants) | 9 | 3 | 3 | 6 | 33
percentage of participants
  Any Paclitaxel-related TEAE | 89 | 100 | 100 | 100 | 94
  Nausea | 33 | 33 | 33 | 50 | 27
  Diarrhea | 33 | 33 | 67 | 50 | 33
  Vomiting | 22 | 0 | 33 | 33 | 24
  Fatigue | 67 | 100 | 33 | 83 | 52
  Edema peripheral | 0 | 0 | 0 | 17 | 15
  Pyrexia | 11 | 0 | 33 | 0 | 15
  Anemia | 67 | 67 | 33 | 33 | 64
  Neutropenia | 22 | 33 | 33 | 33 | 12
  Decreased appetite | 44 | 33 | 0 | 67 | 24
  Hypophosphatemia | 11 | 33 | 0 | 0 | 12
  Alopecia | 11 | 33 | 33 | 67 | 24
  Rash | 11 | 0 | 0 | 0 | 24
  Pruritus | 0 | 33 | 0 | 17 | 12
  Aspartate aminotransferase increased | 0 | 67 | 33 | 33 | 42
  Lymphocyte count decreased | 11 | 0 | 0 | 33 | 36
  White blood cell count decreased | 0 | 67 | 33 | 50 | 33
  Blood creatinine phosphokinase increased | 0 | 33 | 67 | 17 | 6
  Neutrophil count decreased | 0 | 33 | 0 | 17 | 36
  Alanine aminotransferase increased | 0 | 33 | 33 | 17 | 21
  Blood alkaline phosphatase increased | 0 | 33 | 33 | 17 | 12
  Dysgeusia | 11 | 0 | 33 | 50 | 30
  Neuropathy peripheral | 22 | 0 | 33 | 17 | 12

13. Secondary Outcome: Percentage of Participants With PLX3397- and/or Paclitaxel-Related TEAEs (>10%) by Preferred Term (Part 3) (Safety Analysis Set)
Time Frame: From post first dose up to 28 days after the last dose, up to 5 years 9 months
Population: Safety events were assessed in the Safety Analysis Set.
Measure: Number; unit: percentage of participants
Arm/Group | Part 3: PLX3397 600 mg BID | Part 3: Paclitaxel 80 mg/m^2 | Part 3: PLX3397 600 mg BID + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 7 | 5 | 6
percentage of participants
  Any related TEAE | 85.7 | 100 | 100
  Nausea | 57.1 | 40 | 33.3
  Diarrhea | 57.1 | 20 | 50
  Constipation | 0 | 40 | 0
  Vomiting | 0 | 0 | 33.3
  Abdominal distension | 14.3 | 0 | 16.7
  Stomatitis | 0 | 40 | 16.7
  Fatigue | 42.9 | 20 | 83.3
  Chills | 0 | 0 | 50
  Edema peripheral | 14.3 | 20 | 0
  Dysgeusia | 42.9 | 40 | 16.7
  Neuropathy peripheral | 28.6 | 40 | 16.7
  Dizziness | 0 | 0 | 33.3
  Alopecia | 42.9 | 80 | 16.7
  Pruritus | 14.3 | 20 | 16.7
  Myalgia | 0 | 0 | 33.3
  Alanine aminotransferase increased | 14.3 | 20 | 16.7
  Aspartate aminotransferase increased | 14.3 | 20 | 16.7
  Blood bilirubin increased | 14.3 | 0 | 16.7
  Lymphocyte count decreased | 14.3 | 0 | 16.7
  Neutrophil count decreased | 0 | 0 | 33.3
  Decreased appetite | 42.9 | 40 | 16.7
  Anemia | 14.3 | 20 | 33.3
  Neutropenia | 0 | 20 | 16.7

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were recorded from the time the patient received the first dose of study drug up to 28 days after the last dose or before the start of a new anti-tumor therapy, whichever occurred first, up to 5 years 9 months.
Description: All-cause mortality is reported for all patients enrolled in the study. Serious and other (not including serious) adverse events are reported for the Safety Population.
Groups:
- Part 3: PLX3397 600 mg BID: All participants with advanced solid tumors who received PLX3397 600 mg BID as lead-in treatment.
- Part 3: Paclitaxel 80 mg/m^2: All participants with advanced solid tumors who received paclitaxel 80 mg/m^2 intravenous weekly as lead-in treatment.
- Part 3: PLX3397 600 mg BID + Paclitaxel 80 mg/m^2: All participants who received PLX3397 600 mg BID + paclitaxel 80 mg/m^2 intravenous weekly as lead-in treatment.
Arm/Group | Part 1: Cohort 1; 600 mg/Day | Part 1: Cohort 2; 800 mg/Day | Part 1: Cohort 3; 1000 mg/Day | Part 1: Cohort 4; 1200 mg/Day | Part 1 and 2: Cohort 5; 1600 mg/Day | Part 3: PLX3397 600 mg BID | Part 3: Paclitaxel 80 mg/m^2 | Part 3: PLX3397 600 mg BID + Paclitaxel 80 mg/m^2
All-Cause Mortality (participants affected / at risk) | 1/9 | 0/3 | 1/3 | 1/6 | 5/33 | 1/7 | 1/6 | 1/7
Serious Adverse Events (participants affected / at risk) | 1/9 | 1/3 | 3/3 | 2/6 | 10/33 | 5/7 | 2/5 | 3/6
Other Adverse Events (participants affected / at risk) | 9/9 | 3/3 | 3/3 | 6/6 | 33/33 | 7/7 | 5/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Cohort 1; 600 mg/Day (N=9) | Part 1: Cohort 2; 800 mg/Day (N=3) | Part 1: Cohort 3; 1000 mg/Day (N=3) | Part 1: Cohort 4; 1200 mg/Day (N=6) | Part 1 and 2: Cohort 5; 1600 mg/Day (N=33) | Part 3: PLX3397 600 mg BID (N=7) | Part 3: Paclitaxel 80 mg/m^2 (N=5) | Part 3: PLX3397 600 mg BID + Paclitaxel 80 mg/m^2 (N=6)
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device-related sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Puncture site infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal bacteremia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sudden cardiac death (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mixed liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Cohort 1; 600 mg/Day (N=9) | Part 1: Cohort 2; 800 mg/Day (N=3) | Part 1: Cohort 3; 1000 mg/Day (N=3) | Part 1: Cohort 4; 1200 mg/Day (N=6) | Part 1 and 2: Cohort 5; 1600 mg/Day (N=33) | Part 3: PLX3397 600 mg BID (N=7) | Part 3: Paclitaxel 80 mg/m^2 (N=5) | Part 3: PLX3397 600 mg BID + Paclitaxel 80 mg/m^2 (N=6)
Nausea (Gastrointestinal disorders) | 4 | 1 | 2 | 4 | 14 | 5 | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 2 | 3 | 13 | 4 | 2 | 3
Vomiting (Gastrointestinal disorders) | 3 | 0 | 1 | 2 | 12 | 1 | 2 | 3
Constipation (Gastrointestinal disorders) | 3 | 0 | 1 | 0 | 7 | 2 | 3 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 5 | 0 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 2 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 7 | 3 | 1 | 5 | 23 | 3 | 4 | 6
Oedema peripheral (General disorders) | 1 | 1 | 0 | 2 | 9 | 1 | 2 | 0
Pyrexia (General disorders) | 2 | 0 | 1 | 1 | 6 | 0 | 0 | 3
Pain (General disorders) | 1 | 0 | 0 | 0 | 4 | 0 | 1 | 0
Face oedema (General disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Axillary pain (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Feeling jittery (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sudden cardiac death (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 7 | 2 | 1 | 2 | 22 | 2 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 2 | 4 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 1 | 0 | 4 | 12 | 3 | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 2 | 9 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 8 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 4 | 8 | 3 | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 9 | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 5 | 1 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 3 | 11 | 2 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 6 | 1 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 3 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 2 | 1 | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1 | 2 | 14 | 1 | 1 | 1
Lymphocyte count decreased (Investigations) | 1 | 2 | 1 | 2 | 12 | 1 | 0 | 1
Blood creatinine phosphokinase increased (Investigations) | 0 | 1 | 2 | 1 | 13 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 1 | 12 | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 1 | 7 | 1 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 1 | 7 | 0 | 1 | 0
Respiratory rate increased (Investigations) | 0 | 0 | 1 | 1 | 4 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hematocrit decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary physical examination abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 1 | 3 | 12 | 3 | 2 | 2
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 1 | 4 | 2 | 1 | 2
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 1 | 1 | 4 | 2 | 3 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 4 | 1 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 2 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Puncture site infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sialoadenitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 0 | 3 | 10 | 0 | 0 | 3
Systolic hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 1 | 1 | 0 | 5 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 5 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 5 | 1 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye swelling (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 4 | 1 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 5 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sensation of foreign body (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Onychalgia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Percarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mixed liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-03): https://cdn.clinicaltrials.gov/large-docs/02/NCT01525602/Prot_SAP_000.pdf